CLINICAL TRIAL: NCT04136678
Title: The Effect of Treadmill Back Walking Training on Balance and Function in Cerebral Palsy
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, halis dogan, Physiotherapist, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: halisdogan
Record Dates: First submitted 2019-10-10; First posted 2019-10-23 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; treadmill; backward walking; balance; spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Those who are between 6 and 18 years old and have a medical report on the diagnosis of cerebral palsy,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treadmill back walking training (Experimental): 15 minutes conventional walking training, 15 minutes of treadmill back walking training, 15-minute treadmill forward walking training
  Interventions: Other: walking training

INTERVENTIONS:
Other: walking training — 15 minutes of conventional walking training 15 minutes of treadmill backward walking training 15 minutes of treadmil forward walking training
  Other Names: conventional walking training; treadmill backward walking training; treadmill forward walking training

SUMMARY:
The aim of this study was to investigate the effect of treadmill back walking training on balance and function in cerebral palsy.

In our study, scientific data will be prepared by clinical measurement tools in order to determine whether there is balance and walking effect of easy and practicable treadmill back walking training in the clinical setting in Cerebral Palsy.

DETAILED DESCRIPTION:
Measurements will be made at baseline and after each 8 weeks of physiotherapy program, the results will be compared.

30 minutes of the physiotherapy session, which we will apply for 2 days and 45 minutes; in the prone, supine, crawling and above knee positions; They will take physiotherapy training based on neurodevelopmental therapy consisting of fine motor activities, standing up, weight transfer, stretching, strengthening and balance exercises with mat activities such as rotation, weight transfer, sitting.

1. Term: After the first measurements, the participants will take 8 minutes, 2 days a week, the regular physiotherapy session based on 30 minutes Neurodevelopmental Therapy as described above, as well as 15 minutes conventional walking training, then the measurements will be repeated.
2. Term: After the second measurements, the participants will take 8 weeks, 2 days a week, the regular physiotherapy session based on 30 minutes of Neurodevelopmental Therapy as described above, as well as 15 minutes of treadmill back walking training, then the measurements will be repeated.
3. Term: After the third measurements, the participants will take 8 weeks, 2 days a week, the regular physiotherapy session based on the 30 minute Neurodevelopmental Therapy described above, as well as the 15-minute treadmill walking forward training, then the measurements will be repeated.

Statistical method (s) to be used: In the analysis of the results to be obtained in our study, SPS statistics 22.0 version of SPSS statistical package will be used under the Windows operating system Statistical Package for Social Sciences (SPSS). Descriptive statistical information will be shown as arithmetic mean ± Standard Deviation (x statistical ± Ss) or percentage (%) and the level of statistical significance will be considered as p≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Those who are between 6 and 18 years old and have a medical report on the diagnosis of cerebral palsy,
* Classes classified as Level I and II by Gross Motor Function Classification System (GMFCS),
* Lower extremity spasticity classified as 1st and 2nd degree according to Modified Modified Ashworth Scale,
* To understand and apply verbal commands and instructions.
* Volunteer to participate in the study,
* Read and approve the informed consent form.

Exclusion Criteria:

* Active epileptic seizures
* Those with visual or auditory defects,
* Those with fixed deformities in the lower extremities,
* Patients with a history of surgery in the lower extremity musculoskeletal system in the last 6 months
* Injection of Botulinum Toxin (BOTOX) for lower extremity within the last 6 months Spasticity drug users,
* Those with mental and cognitive problems will be excluded from the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
The Pediatric Balance Scale | 8 weeks
  It can be considered as a simple, valid scale for studying functional balance capacity in children with spastic SP (Yi 2012). Pediatric Berg Balance Scale (PBBS) will be used to evaluate the functional balance of daily living activities. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The Rivermead Visual Gait Assessment | 8 weeks
  RVGA allows rapid assessment and documentation of gait disturbances without equipment in the clinic and demonstration of clinical changes (Lord, et al. 1998). Visual parameters of walking in our study will be evaluated by The Rivermead Visual Gait Assessment (RVGA). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: H D Doğan, Pt, Principal Investigator — Istanbul Medipol University Hospital
Locations (1):
- Halkalı, Yükselen Başarı, Abı Hayat, Altın, Özlem and Çocuklarla Elele Education and Rehabilitation Center., Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No